CLINICAL TRIAL: NCT01029639
Title: Effects of Pulsatile Intravenous Insulin Delivery on Hypoglycemic Unawareness
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Administrative
Sponsor: Florida Atlantic University (Other)
Collaborators: Advanced Diabetes Treatment Centers (Other); Global Infusions (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H08-248; MH42900 and MH01386
Record Dates: First submitted 2009-08-06; First posted 2009-12-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Hypoglycemia
Keywords: Pulsatile intravenous insulin; Oral carbohydrate loading; Respiratory Quotients; Hypoglycemia; Diabetes Mellitus, with complications
MeSH Terms: conditions — Hypoglycemia; Diabetes Complications | interventions — Insulin; Insulin Aspart

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (No Intervention): Diabetic patients will complete hypoglycemia unawareness questionnaires at baseline and quarterly thereafter to monitor and assess progress with complications resulting from their diabetes. Comparisons will be performed on low blood sugar incidences reported by subjects requiring heath care intervention other than by the subject themselves.
- Pulsatile Intravenous Insulin Therapy (Humulin R, Novolog) (Experimental): Endocrinologist reviews patient activation after treatment each week and adjust the amounts of insulin and carbohydrates to be given in the next session
  Interventions: Procedure: Pulsatile Intravenous Insulin Therapy (Humulin R, Novolog)

INTERVENTIONS:
Procedure: Pulsatile Intravenous Insulin Therapy (Humulin R, Novolog) — Endocrinologist reviews patient activation after treatment each week and adjust the amounts of insulin and carbohydrates to be given in the next session
  Other Names: Humulin R, Novolog
  Arms: Pulsatile Intravenous Insulin Therapy (Humulin R, Novolog)

SUMMARY:
Hypoglycemic unawareness is a major problem in the treatment of Diabetes Mellitus. Hypoglycemic unawareness is the inability to recognize or sense early symptoms of low blood sugar. This study was instituted to evaluate the effect of Pulsatile intravenous (IV) Insulin on improving or reinstating the diabetics ability to sense or feel the symptoms associated with low blood sugar.

DETAILED DESCRIPTION:
Hypoglycemic Unawareness is the inability for the diabetic patient to sense early symptoms of low blood sugar. Once blood sugar drops too low without the patient's ability to feel the drop urgent treatment may be necessary to prevent further progression This study was instituted to evaluate the effect of Pulsatile IV Insulin on improving the diabetic patients ability to sense and respond to the symptoms associated with falling blood sugars. Anecdotal reports from patients treated with pulsatile IV insulin therapy for other complications suggest that this treatment may show efficacy in patients with hypoglycemic unawareness. Patients who had lost the ability to sense when their blood sugar was dropping dangerously low regained signs and symptoms related to a drop in blood sugar providing them the ability to treat their low blood sugar before experiencing dangerous complications.This study is designed to compare patients with hypoglycemic unawareness who receive pulsatile IV insulin therapy with a control group.Patients will complete a questionnaire at baseline and quarterly thereafter identifying any progress in the signs and symptoms that they may be able to sense with low blood sugar.

Pulsatile IV insulin therapy encourages the glucose metabolism in diabetics to normalize in multiple organs, especially muscle, retina, liver, kidney and nerve endings. The process fundamentally requires the administration of high dose insulin pulses similar to those secreted by non diabetic humans by their pancreas into the surrounding portal circulation. Oral carbohydrates are given simultaneously to augment the process and prevent hypoglycemia. The process is monitored by frequent measuring of glucose levels and respiratory quotients (RQ). RQ is measured by a metabolic cart which determines the ratio VCO2/VO2. This ratio is specific for the fuel used at any one time by the body. The glucose levels are monitored to keep glucose levels appropriate and the RQ determines the need to readjust the infusion protocol in each patient for subsequent insulin infusion sessions. Pulsatile IV insulin therapy is done over 1-hour periods with a 20 to 90 minute rest period between each treatment. Three treatments are given during a patient visit to the center.

Frequent monitoring of RQ is necessary as these levels change rapidly, depending on the fuel being utilized by the body. IV insulin given in pulses shifts metabolism from primarily fatty acid metabolism to primarily glucose metabolism. This shift is reflected by the increase in respiratory quotient. However during rest periods the RQ may fall back to lower levels. Therefore RQs are done at the beginning and at the end of each insulin infusion session in order to appropriately monitor and adjust insulin and carbohydrate loads to reach optimal activation in each session.

The respiratory quotient (RQ) is a measurement of CO2 exhaled and O2 inhaled and is proportionate to the fuel sources being used by the body, primarily the liver over short periods of time. The higher the RQ, the more glucose and less alternative fuel sources are being utilized. Following the RQ change helps determine the effectiveness of physiological insulin administration in increasing anabolic functions in diabetic individuals. By improving the body's glucose metabolism and thereby causing beneficial effects of anabolic factors, the possibility of serious complications can be decreased. In addition the use of oral carbohydrates at the same time along with the physiologic insulin administration stimulates the appropriate gut hormones which augment this effect, a response which cannot be duplicated with intravenous glucose. The purpose of our studies is to determine whether the physiologic administration of insulin along with the augmenting effect of oral carbohydrates will normalize metabolism in diabetic patients and correlate with an improvement in their manifestations of hypoglycemic unawareness in subjects with diabetes.

The RQ is determined by the use of a metabolic cart. Individuals breathe into a mask for 3-5 minutes after a rest period of 20 or more minutes. The ratio of exhaled volume of CO2 to the inhaled volume of O2 is determined as the RQ. The physiologic range is 0.7 to 1.3. Individuals using fat as a primary fuel have a ratio of 0.7, protein or mixed fuels is 0.8-0.9 and carbohydrate is 0.9-1.0. Those taking excessive calories will have RQs higher than 1.05. The amount of intravenous insulin and oral glucose given is determined by the RQ changes during the previous session.

1. Quinones MJ, Nicholas SB, Lyon CJ, Insulin Resistance and The Endothelium, Current Diabetes Reports 5:246-53, 2005.
2. Parrish R, Petersen KF, Mitochondrial Dysfunction and Type 2 Diabetes, Current Diabetes Reports 5:177-183,2005.

ELIGIBILITY:
Inclusion Criteria:

* Up to 400 patients both male and female between the ages of 20 and 90 diagnosed with type 1 or type 2 diabetes mellitus.
* All patients were diagnosed by their endocrinologists as having hypoglycemic unawareness, inability to sense low blood sugars.
* All patients had failed conventional treatment for hypoglycemic unawareness.
* All patients are taking oral agents and/or insulin for diabetic control.
* All patients are under an endocrinologist's supervision for their diabetes management.
* Endocrinologist must assess and approve patient for participation in this study.
* All patients must demonstrate the ability to swallow without difficulty and the ability to commit to the weekly time requirements associated with the study.

Exclusion Criteria:

* Other causes of complications not related to diabetes.
* Lack of intravenous access.
* Pregnancy.
* Alcohol abuse, drug addiction or the use of illegal drugs.
* HIV positive.
* Inability to breathe into machine for respiratory quotients.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Questionnaires completed by subjects at baseline quarterly to assess ability to sense low blood sugar. Tracking incidences requiring outside assistance including paramedics, ER visits and hospitalizations due to low blood sugar incidences. | Every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Betty Tuller, PhD, Principal Investigator — Florida Atlanctic University
Locations (1):
- Florida Atlantic University Center for Complex Systems and Brain Sciences, Boca Raton, Florida, United States

REFERENCES:
- [Background] Quinones MJ, Nicholas SB, Lyon CJ. Insulin resistance and the endothelium. Curr Diab Rep. 2005 Aug;5(4):246-53. doi: 10.1007/s11892-005-0018-z. PMID 16033673